CLINICAL TRIAL: NCT02839785
Title: Analgesia and Physiotherapy in Children With Cerebral Palsy (ANTALKINECP): Double Blind Cross-over Placebo Controlled Study of Ibuprofen in Children With Cerebral Palsy Undergoing Physiotherapy
Brief Title: Analgesia and Physiotherapy in Children With Cerebral Palsy (ANTALKINECP)
Acronym: ANTALKINECP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ANTALKINECP RB15.213
Record Dates: First submitted 2016-06-24; First posted 2016-07-21 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Physiotherapy; Children; Ibuprofen; Pain; Anxiety
MeSH Terms: conditions — Cerebral Palsy; Pain; Anxiety Disorders | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Experimental): Active ibuprofen
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Placebo of ibuprofen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — the child will take orally 30 minutes before each session of physiotherapy 10mg/kg of Ibuprofen (not to exceed 400 mg) in liquid form or placebo.
  Other Names: AdvilMed
  Arms: Ibuprofen
Drug: Placebo — the child will take orally 30 minutes before each session of physiotherapy 10mg/kg of Ibuprofen (not to exceed 400 mg) in liquid form or placebo.
  Arms: Placebo

SUMMARY:
SPARCLE 1 and 2 studies followed a cohort of 818 children with cerebral palsy (CP) between 8 and 12 (SPARCLE 1) and 13 and 18 years old (SPARCLE 2) interviewed at home. The prevalence of pain in these populations was respectively 60 and 69% while it is about 35% in typically developed children of the same age.

The main location of the pain for 60% of children with CP was the lower limbs, caused by musculoskeletal pain and movement (for those who can) and therapeutic procedures. In SPARCLE 2, 50% of the children complained about pain during physical therapy.

If the pain is part of the management of physiotherapy, a recent review showed that for a condition such as chronic back pain, the level of evidence of the effectiveness of physiotherapy techniques in reducing pain is low. The effectiveness of these techniques would include higher efficacy on anxiety than pain itself.

Despite significant involvement of physiotherapists in the management of pain, the focus on pain should increase, in particular taking into account the procedural/induced pain (caused by treatment).

In addition to drugs, physical methods (analgesic therapy) or psychotherapy are used to reduce the pain of children during medical procedures. For the latter most of them require the presence of two individuals to provide the therapy. This is unsuited for out-patient care provided to the majority of children with CP.

Non steroid anti-inflammatory drug (NSAIDs), are first recommended, alone or in combination with the treatment of several indications in child pain (migraine, postoperative pain, etc.). Ibuprofen is commonly used in children during painful procedures and represented the 4th molecule among prescribed per os analgesic drugs in 2008 in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy hemiplegic diplegic or tetraplegic spastic or not.
* Children who feel pain during the pre-screening physiotherapy session with a VAS score above 2.
* Aged 6 to 17 years of both gender.
* Ability to express his/her pain and to measure its intensity with VAS.
* Informed and signed (parents, investigator and child if possible).

Exclusion Criteria:

* Lack of physiotherapy.
* Analgesic treatment already available or stopped in the last month.
* Scheduled surgery procedure or botulinum toxin injection during the period of the assessment of pain (around 5 month)
* The last botulinum toxin injection in two months before the inclusion
* Child who feel pain with EVA score superior or equal to 4 at the time of the inclusion outside the sessions of physiotherapy
* Child unable to cooperate.
* Severe infection or instable vital functions.
* Hypersensitivity to ibuprofen or any of the constituents in the product.
* History of allergy or asthma triggered by taking ibuprofen or substances of near activity such as other NSAIDs and aspirin.
* Allergy to other component of treatment.
* History of upper gastrointestinal bleeding or perforation, related to previous NSAID therapy.
* Active gastrointestinal ulcer.
* Severe hepatic failure.
* Severe renal failure.
* Uncontrolled severe cardiac failure.
* Systemic Lupus Erythematosus.
* Regular intake of ibuprofen

Randomisation Criteria:

• Child who feel pain during the physiotherapy session with a mean VAS score above 3 during the screening phase.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Reduction of at least 20% of the average VAS between the run-in phase and the treatment phase (placebo and ibuprofen) | 5 months

SECONDARY OUTCOMES:
Pain | 5 months
  The pain reduction assessed by the Child health questionnaire
Anxiety | 5 months
  The anxiety reduction assessed by a VAS scale.
Quality of life | 5 months
  The increase in quality of life assessed by the CP Child.
Incidence of adverse events | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Brochard, Dr, Principal Investigator — University hospital of Brest
Locations (3):
- France (3):
  - Hôpital Morvan - CHRU Brest, Brest
  - Hopitaux de Saint-Maurice, Saint-Maurice
  - Ch Lannion-Trestel, Trévou-Tréguignec